CLINICAL TRIAL: NCT04706819
Title: Clinical, Laboratory and Imaging Features, Treatment Trends and Long Term Outcomes in Patients With Parenchymal and Extraparenchymal Neurocysticercosis-A Registry Based Study
Brief Title: Parenchymal and Extraparenchymal Neurocysticercosis-A Registry Based Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Arunmozhimaran Elavarasi, Assistant Professor, Department of Neurology, All India Institute of Medical Sciences
Other Study IDs: IEC-1176/04.12.2020
Record Dates: First submitted 2021-01-03; First posted 2021-01-13 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Neurocysticercosis; Tropical Disease; Tenia Solium Infection
Keywords: Parenchymal Neurocysticercosis; Extraparenchmal Neurocysticercosis; Intraventricular neurocysticercosis; Racemose neurocysticercosis
MeSH Terms: conditions — Neurocysticercosis; Taeniasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Blood and CSF
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Neurocysticercosis(NCC) is the commonest parasitic infection of the central nervous system. It is the commonest cause of focal seizures in India. It can also present with headaches, movement disorders, stroke, cognitive decline and multitude of complications depending on its location. Parenchymal NCC is more common than extraparenchymal NCC. There is considerable variation in the treatment practices including administration of anti-helminthic agents and corticosteroids. Extra-parenchymal NCC is rare and can occur in the subarachnoid space or intraventricularly. Extra-parenchymal NCC is managed surgically in several instances. There is scant literature on the long term follow up of this condition. This registry will enable collection of data on the clinical, laboratory and imaging features, treatment trends and long term outcomes of both parenchymal and extra-parenchymal neurocysticercosis.

DETAILED DESCRIPTION:
Neurocysticercosis (NCC) is the commonest parasitic infection of the central nervous system. It can affect the brain, meninges, eyes as well as other parts of the body. Disseminated cysticercosis involves brain and one other organ such as muscles, viscera etc. NCC is common in tropical countries and is the commonest cause of focal seizures. It is quite frequently also found incidentally in imaging done for unrelated conditions such as headaches and trauma. NCC can be parenchymal or extra-parenchymal. Parenchymal NCC is commoner than extra-parenchymal lesions. Some patients with parenchymal NCC have less than three cysts and they have seizures which are well controlled with medication. On the other hand some have multiple cysts and present with complications such as stroke, cognitive decline, aphasia, hydrocephalus, increased intra-cranial pressure etc. Cysts occurring extra-parenchymal locations such as inside the ventricular system or sub-arachnoid space are less common than parenchymal ones, but can be more symptomatic due to obstruction in the CSF flow leading to hydrocephalus, arachnoiditis and impaired CSF absorption etc.

Though NCC is very common in the Indian subcontinent, there is no consensus on optimum management strategies. There is a wide variation in the practices of prescribing anti-helminthic drugs, corticosteroids, steroid sparing agents etc. Clinical experience suggests that some patients with NCC need long term corticosteroids and on withdrawing corticosteroids, they develop peri-lesional edema and they become symptomatic. In such patients, steroid sparing agents such as methotrexate are recommended.2 However there is no data on the long term follow up of such patients especially from India. Similarly, patients with intraventricular NCC treated surgically are given varying types of anti-helminthic therapy ranging from none to combination therapy after surgical /endoscopic resection of the cysts.

It is high time, that a registry is established and patient data collected systematically, to enable analysis of clinical features as well as to study the patterns of treatment offered by individual physicians. This will also promote the development of hypothesis for planning trials in future.

ELIGIBILITY:
Inclusion Criteria:

* Patients attending Neurology OPD or are admitted in wards with neurocysticercosis diagnosed on the basis of composite clinical criteria, imaging criteria as well as natural history
* Atleast 14 years of age of all sexes
* Reasonable clinical certainty OR allied investigations such as CXR/CECT chest/abdomen/PET CT as per clinical indication ruling out tuberculosis or mimics of neurocysticercosis
* Other relevant investigations like CSF analysis not suggestive of alternative diagnosis such as tubercular/ cryptococcal/other fungal infections/other causes of chronic meningitis such as brucella/ nocardia/ syphilis/recurrent viral meningitis/ carcinomatous/ lymphomatous meningitis or non infective causes such as sarcoidosis/sub-arachnoid hemorrhage etc.

Exclusion Criteria:

• Not willing to provide consent

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study Population: Patients with MRI/CT diagnosed neurocysticercosis as per composite clinical criteria, imaging criteria as well as natural history
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-01-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical features in patients with parenchymal and extraparenchymal neurocysticercosis | 6 months
  To study the clinical features in patients with parenchymal and extraparenchymal neurocysticercosis
Laboratory features | 6 months
  To study the hematologic and CSF parameters in patients with parenchymal and extraparenchymal neurocysticercosis
Imaging features | 6 months
  To study the imaging features in patients with parenchymal and extraparenchymal neurocysticercosis
Treatment trends in patients with parenchymal and extraparenchymal neurocysticercosis | 6 months
  To study the treatment trends in terms of proportion of patients treated with anti-epileptic drugs, anti-parasitic drugs, corticosteroids, steroid sparing agents, surgical management in patients with parenchymal and extraparenchymal neurocysticercosis
Treatment trends in patients with parenchymal and extraparenchymal neurocysticercosis | 1 year
  To study the treatment trends in terms of proportion of patients treated with anti-epileptic drugs, anti-parasitic drugs, corticosteroids, steroid sparing agents, surgical management in patients with parenchymal and extraparenchymal neurocysticercosis
Treatment trends in patients with parenchymal and extraparenchymal neurocysticercosis | 3 years
  To study the treatment trends in terms of proportion of patients treated with anti-epileptic drugs, anti-parasitic drugs, corticosteroids, steroid sparing agents, surgical management in patients with parenchymal and extraparenchymal neurocysticercosis
Treatment trends in patients with parenchymal and extraparenchymal neurocysticercosis | 5 years
  To study the treatment trends in terms of proportion of patients treated with anti-epileptic drugs, anti-parasitic drugs, corticosteroids, steroid sparing agents, surgical management in patients with parenchymal and extraparenchymal neurocysticercosis
Outcomes in patients with parenchymal and extraparenchymal neurocysticercosis - 6 months | 6 months
  To study the outcomes in terms of seizure freedom, symptom resolution, new symptoms, imaging resolution and functional status in patients with parenchymal and extraparenchymal neurocysticercosis
Outcomes in patients with parenchymal and extraparenchymal neurocysticercosis | 1 year
  To study the outcomes in terms of seizure freedom, symptom resolution, new symptoms, imaging resolution and functional status in patients with parenchymal and extraparenchymal neurocysticercosis
Outcomes in patients with parenchymal and extraparenchymal neurocysticercosis | 3 years
  To study the outcomes in terms of seizure freedom, symptom resolution, new symptoms, imaging resolution and functional status in patients with parenchymal and extraparenchymal neurocysticercosis
Outcomes in patients with parenchymal and extraparenchymal neurocysticercosis | 5 years
  To study the outcomes in terms of seizure freedom, symptom resolution, new symptoms, imaging resolution and functional status in patients with parenchymal and extraparenchymal neurocysticercosis
Extra-parenchymal neurocysticercosis | 6 months
  To find the proportion of patients having extra-parenchymal neurocysticercosis

SECONDARY OUTCOMES:
Factors determining outcomes in patients with parenchymal neurocysticercosis | 1 year
  To study the factors determining outcomes in terms of seizure freedom, resolution of symptoms, disappearance of lesions on imaging and functional status as assessed by modified Rankin scale in patients with parenchymal neurocysticercosis
Factors determining outcomes in patients with parenchymal neurocysticercosis | 3 years
  To study the factors determining outcomes in terms of seizure freedom, resolution of symptoms, disappearance of lesions on imaging and functional status as assessed by modified Rankin scale in patients with parenchymal neurocysticercosis
Factors determining outcomes in patients with parenchymal neurocysticercosis | 5 years
  To study the factors determining outcomes in terms of seizure freedom, resolution of symptoms, disappearance of lesions on imaging and functional status as assessed by modified Rankin scale in patients with parenchymal neurocysticercosis
Factors determining outcomes in patients with extra-parenchymal neurocysticercosis | 1 year
  To study the factors determining outcomes in terms of seizure freedom, resolution of symptoms, disappearance of lesions on imaging and functional status as assessed by modified Rankin scale in patients with extra-parenchymal neurocysticercosis
Factors determining outcomes in patients with extra-parenchymal neurocysticercosis | 5 years
  To study the factors determining outcomes in terms of seizure freedom, resolution of symptoms, disappearance of lesions on imaging and functional status as assessed by modified Rankin scale in patients with extra-parenchymal neurocysticercosis

CONTACTS AND LOCATIONS:
Overall Officials: Arunmozhimaran Elavarasi, MD DM, Principal Investigator — All India Institute of Medical Sciences; Ajay Garg, MD DM, Principal Investigator — All India Institute of Medical Sciences

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Garcia HH, Nash TE, Del Brutto OH. Clinical symptoms, diagnosis, and treatment of neurocysticercosis. Lancet Neurol. 2014 Dec;13(12):1202-15. doi: 10.1016/S1474-4422(14)70094-8. Epub 2014 Nov 10. PMID 25453460
- [Background] White AC Jr, Coyle CM, Rajshekhar V, Singh G, Hauser WA, Mohanty A, Garcia HH, Nash TE. Diagnosis and Treatment of Neurocysticercosis: 2017 Clinical Practice Guidelines by the Infectious Diseases Society of America (IDSA) and the American Society of Tropical Medicine and Hygiene (ASTMH). Clin Infect Dis. 2018 Apr 3;66(8):e49-e75. doi: 10.1093/cid/cix1084. No abstract available. PMID 29481580
- [Background] Rajshekhar V. Evolution of concepts in the management of cysticercosis of the brain: Then (1970) and now (2018). Neurol India. 2018 Jul-Aug;66(4):919-927. doi: 10.4103/0028-3886.236969. No abstract available. PMID 30038069
- [Background] Rajshekhar V, Raghava MV, Prabhakaran V, Oommen A, Muliyil J. Active epilepsy as an index of burden of neurocysticercosis in Vellore district, India. Neurology. 2006 Dec 26;67(12):2135-9. doi: 10.1212/01.wnl.0000249113.11824.64. PMID 17190933
- [Background] Moyano LM, Saito M, Montano SM, Gonzalvez G, Olaya S, Ayvar V, Gonzalez I, Larrauri L, Tsang VC, Llanos F, Rodriguez S, Gonzalez AE, Gilman RH, Garcia HH; Cysticercosis Working Group in Peru. Neurocysticercosis as a cause of epilepsy and seizures in two community-based studies in a cysticercosis-endemic region in Peru. PLoS Negl Trop Dis. 2014 Feb 13;8(2):e2692. doi: 10.1371/journal.pntd.0002692. eCollection 2014 Feb. PMID 24551255
- [Background] Garcia HH, Gonzales I, Lescano AG, Bustos JA, Zimic M, Escalante D, Saavedra H, Gavidia M, Rodriguez L, Najar E, Umeres H, Pretell EJ; Cysticercosis Working Group in Peru. Efficacy of combined antiparasitic therapy with praziquantel and albendazole for neurocysticercosis: a double-blind, randomised controlled trial. Lancet Infect Dis. 2014 Aug;14(8):687-695. doi: 10.1016/S1473-3099(14)70779-0. Epub 2014 Jul 3. PMID 24999157
- [Background] Nash TE, Pretell EJ, Lescano AG, Bustos JA, Gilman RH, Gonzalez AE, Garcia HH; Cysticercosis Working Group in Peru. Perilesional brain oedema and seizure activity in patients with calcified neurocysticercosis: a prospective cohort and nested case-control study. Lancet Neurol. 2008 Dec;7(12):1099-105. doi: 10.1016/S1474-4422(08)70243-6. Epub 2008 Nov 3. PMID 18986841
- [Background] Ooi WW, Wijemanne S, Thomas CB, Quezado M, Brown CR, Nash TE. Short report: A calcified Taenia solium granuloma associated with recurrent perilesional edema causing refractory seizures: histopathological features. Am J Trop Med Hyg. 2011 Sep;85(3):460-3. doi: 10.4269/ajtmh.2011.11-0221. PMID 21896805
- [Background] Sheth TN, Pillon L, Keystone J, Kucharczyk W. Persistent MR contrast enhancement of calcified neurocysticercosis lesions. AJNR Am J Neuroradiol. 1998 Jan;19(1):79-82. PMID 9432161
- [Background] Amaral L, Maschietto M, Maschietto R, Cury R, Ferreira NF, Mendonca R, Lima SS. Ununsual manifestations of neurocysticercosis in MR imaging: analysis of 172 cases. Arq Neuropsiquiatr. 2003 Sep;61(3A):533-41. doi: 10.1590/s0004-282x2003000400002. Epub 2003 Sep 16. PMID 14513153
- [Background] Huang X, Wang Z, Kou J, Liu H, Mao D, Yu Z, Liu X, Cheng P, Gong M. A Large Cohort of Neurocysticercosis in Shandong Province, Eastern China, 1997-2015. Vector Borne Zoonotic Dis. 2019 Dec;19(12):901-907. doi: 10.1089/vbz.2019.2447. Epub 2019 Jul 17. PMID 31314709
- [Background] Martinez HR, Rangel-Guerra R, Elizondo G, Gonzalez J, Todd LE, Ancer J, Prakash SS. MR imaging in neurocysticercosis: a study of 56 cases. AJNR Am J Neuroradiol. 1989 Sep-Oct;10(5):1011-9. PMID 2505513
- [Background] Abba K, Ramaratnam S, Ranganathan LN. Anthelmintics for people with neurocysticercosis. Cochrane Database Syst Rev. 2010 Jan 20;(1):CD000215. doi: 10.1002/14651858.CD000215.pub3. PMID 20091504
- [Background] Garcia HH, Pretell EJ, Gilman RH, Martinez SM, Moulton LH, Del Brutto OH, Herrera G, Evans CA, Gonzalez AE; Cysticercosis Working Group in Peru. A trial of antiparasitic treatment to reduce the rate of seizures due to cerebral cysticercosis. N Engl J Med. 2004 Jan 15;350(3):249-58. doi: 10.1056/NEJMoa031294. PMID 14724304
- [Background] Nash TE, Ware JM, Mahanty S. Intraventricular Neurocysticercosis: Experience and Long-Term Outcome from a Tertiary Referral Center in the United States. Am J Trop Med Hyg. 2018 Jun;98(6):1755-1762. doi: 10.4269/ajtmh.18-0085. Epub 2018 Apr 19. PMID 29692305
- [Background] Sinha S, Sharma BS. Intraventricular neurocysticercosis: a review of current status and management issues. Br J Neurosurg. 2012 Jun;26(3):305-9. doi: 10.3109/02688697.2011.635820. Epub 2011 Dec 15. PMID 22168964
- [Background] Suri A, Goel RK, Ahmad FU, Vellimana AK, Sharma BS, Mahapatra AK. Endoscopic excision of intraventricular neurocysticercosis in children: a series of six cases and review. Childs Nerv Syst. 2008 Feb;24(2):281-5. doi: 10.1007/s00381-007-0462-y. Epub 2007 Nov 10. PMID 17994242
- [Background] Suri A, Goel RK, Ahmad FU, Vellimana AK, Sharma BS, Mahapatra AK. Transventricular, transaqueductal scope-in-scope endoscopic excision of fourth ventricular neurocysticercosis: a series of 13 cases and a review. J Neurosurg Pediatr. 2008 Jan;1(1):35-9. doi: 10.3171/PED-08/01/035. PMID 18352801
- [Background] Sharma BS, Sawarkar DP, Verma SK. Endoscopic Management of Fourth Ventricle Neurocysticercosis: Description of the New Technique in a Case Series of 5 Cases and Review of the Literature. World Neurosurg. 2019 Feb;122:e647-e654. doi: 10.1016/j.wneu.2018.10.117. Epub 2018 Oct 26. PMID 30814022
- [Background] Proano JV, Torres-Corzo J, Rodriguez-Della Vecchia R, Guizar-Sahagun G, Rangel-Castilla L. Intraventricular and subarachnoid basal cisterns neurocysticercosis: a comparative study between traditional treatment versus neuroendoscopic surgery. Childs Nerv Syst. 2009 Nov;25(11):1467-75. doi: 10.1007/s00381-009-0933-4. Epub 2009 Jun 26. PMID 19557421
- [Background] Nash TE, O'Connell EM, Hammoud DA, Wetzler L, Ware JM, Mahanty S. Natural History of Treated Subarachnoid Neurocysticercosis. Am J Trop Med Hyg. 2020 Jan;102(1):78-89. doi: 10.4269/ajtmh.19-0436. PMID 31642423